CLINICAL TRIAL: NCT02583165
Title: A Phase 1 Study of MEDI1873 (GITR Agonist) in Adult Subjects With Select Advanced Solid Tumors
Brief Title: A Study in Adult Subjects With Select Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6150C00001
Record Dates: First submitted 2015-10-19; First posted 2015-10-22 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; immunotherapy; immuno-oncology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monotherapy arm (Experimental): MEDI1873
  Interventions: Biological: MEDI1873

INTERVENTIONS:
Biological: MEDI1873 — Subjects will receive MEDI1873 by intravenous administration

SUMMARY:
To evaluate the safety and tolerability of MEDI1873 in adult subjects with selected advanced solid tumors.

DETAILED DESCRIPTION:
This is a first-time-in-human, Phase 1, multicenter, open-label, single-arm dose-escalation study of MEDI1873 to evaluate the safety, tolerability, pharmacokinetics, immunogenicity, pharmacodynamics and anti-tumor activity in adult subjects with advanced solid tumor malignancies

ELIGIBILITY:
Inclusion Criteria:

* All subjects must consent to provide archived tumor specimen
* Subjects must have histologically or cytologically confirmed advanced solid tumor for recurrent or metastatic disease.
* At the time of Day 1 of the study, subjects with central nervous system (CNS) metastases must have been treated and must be asymptomatic
* Willingness to provide pretreatment and on-treatment biopsies.
* Adequate organ function
* Females of childbearing potential and nonsterilized males who are sexually active must use effective methods of contraception

Exclusion Criteria:

* Known allergic reaction to any component of MEDI1873
* Concurrent enrollment in another clinical study, unless it is an observational clinical study or the follow-up period of an interventional study
* Receipt of any anticancer therapy within 4 weeks prior to the first dose of MEDI1873; in the case of mAbs, 6 weeks prior to the first dose of MEDI1873
* Any concurrent chemotherapy, immunotherapy, biologic, or hormonal therapy for cancer treatment.
* Receipt of live, attenuated vaccine within 28 days prior to the first dose of investigational product
* Unresolved toxicities from prior anticancer therapy
* Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects with adverse events (AEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs) | From time of informed consent through 12 months after last dose of MEDI1873
  The maximum tolerated dose (MTD)/highest protocol-defined dose level in the absence of establishing an MTD will be determined by the number of participants experiencing DLTs. The safety profile will be assessed through number of participants experiencing AEs, SAEs, DLTs, abnormal laboratory parameters, vital signs and electrocardiogram (ECG) results.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated to be from time of informed consent up to 4.5 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Disease control rate (DCR) | Estimated to be from time of informed consent up to 4.5 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1
Duration of response (DoR) | Estimated to be from time of informed consent up to 4.5 years
  Duration of response will be defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Estimated to be from time of informed consent up to 4.5 years
  Progression-free survival will be measured from the start of treatment with MEDI1873 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Estimated to be from time of informed consent up to 4.5 years
  Overall survival will be determined as the time from the start of treatment with MEDI1873 until death due to any cause.
Maximum observed concentration (Cmax) of MEDI1873 | From first dose of MEDI1873 through to 30 days after last dose of MEDI1873
  The endpoint for assessment of PK of MEDI1873 include serum concentrations of MEDI1873 at different timepoints after MEDI1873 administration
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of MEDI1873 through to 12 months after last dose of MEDI1873
  The immunogenicity of MEDI1873 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs)
PD biomarkers including changes from baseline levels in various lymphocyte populations | From time of informed consent through to disease progression, assessed up to 4.5 years
  PD biomarkers including changes from baseline levels in various lymphocyte populations
Area under the curve (AUC) of MEDI1873 | From first dose of MEDI1873 through to 30 days after last dose of MEDI1873
  The endpoint for assessment of PK of MEDI1873 include serum concentrations of MEDI1873 at different timepoints after MEDI1873 administration
Clearance (CL) of MEDI1873 | From first dose of MEDI1873 through to 30 days after last dose of MEDI1873
  The endpoint for assessment of PK of MEDI1873 include serum concentrations of MEDI1873 at different timepoints after MEDI1873 administration
Terminal half-life of MEDI1873 | From first dose of MEDI1873 through to 30 days after last dose of MEDI1873
  The endpoint for assessment of PK of MEDI1873 include serum concentrations of MEDI1873 at different timepoints after MEDI1873 administration
Percentage of subjects who develop detectable anti-drug antibodies (ADAs) | From first dose of MEDI1873 through to 12 months after last dose of MEDI1873
  The immunogenicity of MEDI1873 will be assessed by summarizing the percentage of subjects who develop detectable anti-drug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Overall Officials: Medimmune LLC, Study Director — MedImmune LLC
Locations (10):
- United States (10):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, Tampa, Florida
  - Research Site, Rochester, Minnesota
  - Research Site, New York, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas